CLINICAL TRIAL: NCT04059783
Title: Non-interventional Study on the Onset of Effect of Iberogast in Patients With Functional or Motility-related Gastrointestinal Diseases
Brief Title: Study to Learn More About the Onset of Effect of Iberogast in Patients Suffering From Abnormal Stomach and Intestine Function
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20984
Record Dates: First submitted 2019-07-12; First posted 2019-08-16 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — iberogast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: STW5 (Iberogast®, BAY98-7411) — The medication was applied 3 x 20 drops per day orally, before or at meals with some liquid, ideally three weeks

SUMMARY:
Several studies have been done on the efficacy of the herbal medicine Iberogast. In this study researcher want to learn more about the time needed for Iberogast to start to work after the patient took the drug. This study plans to enroll 300 adult male and female patients suffering from disturbance of stomach and intestine normal function and treated by their doctor with Iberogast drops. Patients will be asked to document on a diary card the changes of symptom severity of the stomach and intestine complaints and the time needed for the symptoms to improve after drug intake. At the end of the study the treating doctor and the patients will be asked about the overall changes of symptoms. In addition information on the safety of the drug and how well the drug is tolerated by the patients will be collected

ELIGIBILITY:
Inclusion criteria:

At the discretion of physician under the instructions of Rome III criteria concerning functional gastrointestinal symptoms as well as the summary of product characteristics of Iberogast

Exclusion criteria:

Therapeutic necessity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients of at least 18 years were to be observed
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2008-06-17 (Actual); Primary Completion 2010-04-27 (Actual); Study Completion 2011-02-20 (Actual)

PRIMARY OUTCOMES:
Change of GIS score from baseline up to 3 weeks after treatment | At baseline and up to 3 weeks post-treatment
  Gastrointestinal System Profile (GIS) includes 5 scores: 0=Not available, 1=Slight, 2=Moderate, 3=Severe, 4=Very severe
Global assessment by the physicians using a 4-point likert scale | Up to 3 weeks
  Therapeutic success assessed by physicians. 0=Not improved, 1=Slightly improved, 2=Significantly approved, 3=No symptoms
Global assessment by the patient using a 4-point likert scale | Up to 3 weeks
  Therapeutic success assessed by patient. 0=Not improved, 1=Slightly improved, 2=Significantly approved, 3=No symptoms
Change of ratings of symptom severity on a 100-mm visual analogue scale (VAS) over time after intake of Iberogast | At baseline and up to 2 hours post-treatment on day 1
  Visual Analogue Scale to evaluate the general severity of symptoms. It is an unmarked scale on a line 100 mm in length, indicating from 0 mm (no symptoms) to 100 mm (severe symptoms).
Onset of improvement assessed by patient on day 1 | On day 1
  The onset of effect (severity of the functional gastrointestinal symptoms as well as the time frame within which the symptoms improved) was documented by the patients in the patient diary card. According to the time frame stated in the card (1 minute, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, more than 2 hours), the patients had to mark the time with a cross at which their symptoms significantly improved (i.e. perceived by the patient) following the one-time intake of Iberogast at morning, noon and evening on day 1
Onset of improvement assessed by patient on day 2 | On day 2
  The onset of effect (severity of the functional gastrointestinal symptoms as well as the time frame within which the symptoms improved) was documented by the patients in the patient diary card. According to the time frame stated in the card (1 minute, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, more than 2 hours), the patients had to mark the time with a cross at which their symptoms significantly improved (i.e. perceived by the patient) following the one-time intake of Iberogast at morning, noon and evening on day 2
Onset of improvement assessed by patient on day 3 | On day 3
  The onset of effect (severity of the functional gastrointestinal symptoms as well as the time frame within which the symptoms improved) was documented by the patients in the patient diary card. According to the time frame stated in the card (1 minute, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, more than 2 hours), the patients had to mark the time with a cross at which their symptoms significantly improved (i.e. perceived by the patient) following the one-time intake of Iberogast at morning, noon and evening on day 3
Onset of improvement assessed by patient on day 4 | On day 4
  The onset of effect (severity of the functional gastrointestinal symptoms as well as the time frame within which the symptoms improved) was documented by the patients in the patient diary card. According to the time frame stated in the card (1 minute, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, more than 2 hours), the patients had to mark the time with a cross at which their symptoms significantly improved (i.e. perceived by the patient) following the one-time intake of Iberogast at morning, noon and evening on day 4
Onset of improvement assessed by patient on day 5 | On day 5
  The onset of effect (severity of the functional gastrointestinal symptoms as well as the time frame within which the symptoms improved) was documented by the patients in the patient diary card. According to the time frame stated in the card (1 minute, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, more than 2 hours), the patients had to mark the time with a cross at which their symptoms significantly improved (i.e. perceived by the patient) following the one-time intake of Iberogast at morning, noon and evening on day 5
Onset of improvement assessed by patient on day 6 | On day 6
  The onset of effect (severity of the functional gastrointestinal symptoms as well as the time frame within which the symptoms improved) was documented by the patients in the patient diary card. According to the time frame stated in the card (1 minute, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, more than 2 hours), the patients had to mark the time with a cross at which their symptoms significantly improved (i.e. perceived by the patient) following the one-time intake of Iberogast at morning, noon and evening on day 6
Onset of improvement assessed by patient on day 7 | On day 7
  The onset of effect (severity of the functional gastrointestinal symptoms as well as the time frame within which the symptoms improved) was documented by the patients in the patient diary card. According to the time frame stated in the card (1 minute, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, more than 2 hours), the patients had to mark the time with a cross at which their symptoms significantly improved (i.e. perceived by the patient) following the one-time intake of Iberogast at morning, noon and evening on day 7
Onset of improvement assessed by patient on day 8 | On day 8
  The onset of effect (severity of the functional gastrointestinal symptoms as well as the time frame within which the symptoms improved) was documented by the patients in the patient diary card. According to the time frame stated in the card (1 minute, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, more than 2 hours), the patients had to mark the time with a cross at which their symptoms significantly improved (i.e. perceived by the patient) following the one-time intake of Iberogast at morning, noon and evening on day 8

SECONDARY OUTCOMES:
The number of participants with adverse events | Up to 3 weeks
  Participants who had adverse events during the study
The number of participants who discontinued from treatment | Up to 3 weeks
  Participants who discontinued from study treatment
The number of participants with the need of further treatment | Up to 3 weeks
  Participants who needed further treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/